CLINICAL TRIAL: NCT00369733
Title: Disease/Case Management of Patients Receiving ARANESP™ (Darbepoetin Alfa) to Treat the Anemia of Chronic Renal Insufficiency (CRI)
Brief Title: STAAR-3 Clinical Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Global Development Leader, Amgen Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20010243
Record Dates: First submitted 2006-08-24; First posted 2006-08-29 (Estimated); Last update posted 2010-02-19 (Estimated); Status verified 2010-02

CONDITIONS: Chronic Kidney Disease; Chronic Renal Insufficiency; Kidney Disease; Pre-dialysis; Pre-ESRD
Keywords: Aranesp; Anemia; Kidney Disease; Hemoglobin; darbepoetin alfa; QoL
MeSH Terms: conditions — Renal Insufficiency, Chronic; Kidney Diseases; Anemia | interventions — Darbepoetin alfa

ARMS (1):
- Single arm (Experimental): Aranesp adminsitered every other week for 52 weeks
  Interventions: Drug: Darbepoetin alfa

INTERVENTIONS:
Drug: Darbepoetin alfa — Darbepoetin alfa adminstered SC every other week to acheive a Hb not to exceed 12 g/dL
  Other Names: Aranesp

SUMMARY:
To assess the effect of Aranesp on the hemoglobin (Hgb) of CRI subjects who are recombinant human erythropoietin (rHuEPO)-naïve or converting from rHuEPO therapy.

DETAILED DESCRIPTION:
To assess the effect of Aranesp on the hemoglobin of CRI subjectswho are recombinant human erythropoetin (rHuEPO)-naïve or converting from rHuEPO therapy and to assess the association between subject self-reported health-related quality of life (HRQoL) as it relates to Hgb concentration and glomerular filtration rate (GFR) in subjects who were rHuEPO-naïve prior to study enrollment.

To characterize the health-related resource utilization of subjects with CRI. To characterize the subject satisfaction with Aranesp™ compared to previous rHuEPO therapy.

To characterize iron treatment in subjects with CRI. To evaluate the extent to which implementation of case management contributes to achieving the desired clinical objectives.

To assess the safety profile of Aranesp™ therapy in subjects with CRI.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of CRI and not receiving dialysis therapy (must be predialysis)
* measured or estimated (using the Cockcroft-Gault formula) creatinine clearance (CrCl) of ≤ 70 mL/min, or GFR ≤ 60 mL/min (using the MDRD formula):
* Cockcroft-Gault formula: CrCl = (140 minus age in years) x (body weight in kg) serum creatinine (mg/dL) x 72.0. For women, the value will be multiplied by 0.85
* MDRD formula: GFR = 170 x [SCr]-0.999 x [Age]-0.167 x [0.762 if subject is female] x [1.180 if subject is black] x [SUN]-0.170 x [SAlb]-0.318
* (if subject is not already receiving rHuEPO therapy) mean Hgb < 11 g/dL during the screening/baseline period
* for subjects currently receiving rHuEPO therapy, the subject must have: a stable rHuEPO dose for the past month; and a rHuEPO frequency of once weekly.
* white blood cell and platelet counts within normal limits
* serum vitamin B12 and folate levels above the lower limit of normal range
* transferrin saturation (TSAT) ≥ 20% during the screening period
* availability for follow-up assessments
* subject must be able to comprehend and be willing to, or have legally accepted representative, give written informed consent for participation in the study

Exclusion Criteria:

* scheduled to initiate dialysis
* uncontrolled hypertension (diastolic blood pressure > 105 mm Hg or systolic blood pressure of > 180 mm Hg during the screening/baseline period on two separate measurements)
* clinically unstable in the judgment of the investigator (eg, subject is in the intensive care unit, immediately post-myocardial infarction, etc)
* scheduled to receive a living donor kidney transplant
* treatment of grand mal epilepsy within the past 6 months
* moderate to severe congestive heart failure (NYHA class III or IV)
* clinical evidence of severe secondary hyperparathyroidism (parathyroid hormone level > 1500 pg/mL)
* severe active chronic inflammatory process (eg, ulcerative colitis, peptic ulcer disease, rheumatoid arthritis, etc)
* currently receiving antibiotic therapy for systemic infection (enrollment may be postponed until the course of antibiotics has ended)
* known aspartate aminotransferase (AST) or alanine aminitransferase (ALT) greater than 3 times the upper limit of the normal range on more than one occasion within three months prior to screening
* known positive HIV antibody or hepatitis B surface antigen
* clinical evidence of current malignancy and/or receiving chemotherapy with the exception of basal cell or squamous cell carcinoma of the skin and cervical intraepithelial neoplasia
* active bleeding or RBC transfusion within eight weeks of enrollment
* androgen therapy within four weeks before enrollment
* known hematologic disease (eg, sickle cell anemia, myelodysplastic syndromes, hematologic malignancy, myeloma; hemolytic anemia, etc)
* any condition that is likely to affect subject compliance
* currently or previously (within 30 days) enrolled in investigational device or drug trial(s) or receiving investigational agent(s)
* the exception to this is if the subject was enrolled in another Aranesp™ or rHuEPO protocol
* pregnant or breast feeding women (women of child-bearing potential must be using contraceptive precautions)
* women planning to have a child during the study period
* known hypersensitivity to the active substance or any of the excipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 443 (Actual)
Dates: Start 2002-05; Primary Completion 2004-03 (Actual); Study Completion 2004-05 (Actual)

PRIMARY OUTCOMES:
Mean hemoglobin during the evaluation period. | 52 weeks

SECONDARY OUTCOMES:
Change in hemoglobin throughout the study | 52 weeks
HRQoL scores of rHuEPO-naïve subjects measured at baseline, week 12, week 24, and end of study | 52 weeks
Health-related resource utilization, measured every 4 weeks, throughout the study | 52 weeks
Patient satisfaction scores of subjects previously on rHuEPO therapy, measured at baseline and week 12 | 12 weeks
Iron requirement (dose, frequency, and route) of subjects during the study | 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Derived] Abu-Alfa AK, Sloan L, Charytan C, Sekkarie M, Scarlata D, Globe D, Audhya P. The association of darbepoetin alfa with hemoglobin and health-related quality of life in patients with chronic kidney disease not receiving dialysis. Curr Med Res Opin. 2008 Apr;24(4):1091-100. doi: 10.1185/030079908x280653. Epub 2008 Mar 6. PMID 18328118
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com